CLINICAL TRIAL: NCT05527691
Title: Testing SupportGroove: a Novel Mhealth Intervention for Couples Coping with Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: McGuire Research Institute (Other)
Responsible Party: Principal Investigator, Alexandra Terrill, Associate Professor, Occupational Recreational Therapy, University of Utah
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 720484
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Spinal Cord Injuries; Relationship, Marital
Keywords: spinal cord injuries; couple; relationship; resilience
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SupportGroove (Experimental): 8-week intervention that is remotely delivered through a mobile app, consisting of daily "quests" (positive psychology-based activities) completed individually and as a couple.
  Interventions: Behavioral: SupportGroove
- Waitlist control (No Intervention): Participants will be waitlisted for 8 weeks.

INTERVENTIONS:
Behavioral: SupportGroove — An app-delivered program consisting of positive psychology-based activities, such as expressing gratitude, finding meaning, savoring, and fostering connections. Participants complete daily "quests" suggested through the app, some of which are completed on their own, and some with their partner.
  Arms: SupportGroove

SUMMARY:
The purpose of this study is to test the preliminary effects of an 8-week mobile application-based program (SupportGroove) developed for persons with spinal cord injury and their romantic partners.

DETAILED DESCRIPTION:
Eligible couples who provide informed consent will be enrolled in the study and will be randomized to either immediately start the 8-week SupportGroove program or be waitlisted for 8-weeks before starting the program. While actively participating in the program, couples will use the app to engage in daily "quests" (positive psychology-based activities to be completed on their own or as a couple). Both partners in the participating couple complete self-report assessments at baseline (0 weeks), 8 weeks, 16 weeks, and 28 weeks.

ELIGIBILITY:
Inclusion Criteria:

* cohabitating romantic couples where one partner has sustained a spinal cord injury at least 3 months prior to enrolling in the study
* be able to read and understand printed English instructions
* have a smartphone, tablet, or personal computer with internet access

Exclusion Criteria:

* the partner has a spinal cord injury or other major neurological condition
* either partner is unable to read and understand printed English instructions
* either partner does not consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Spinal Cord Injury Quality of Life (SCI-QOL) Resilience-Short Form | Baseline (0 weeks)
  10-items assessing state resilience; rated from 1-5 (never-always); score range from 19-50, higher score = more resilient /better outcome
Spinal Cord Injury Quality of Life (SCI-QOL) Resilience-Short Form | 8 weeks
  10-items assessing state resilience; rated from 1-5 (never-always); score range from 19-50, higher score = more resilient /better outcome
Spinal Cord Injury Quality of Life (SCI-QOL) Resilience-Short Form | 16 weeks
  10-items assessing state resilience; rated from 1-5 (never-always); score range from 19-50, higher score = more resilient /better outcome
Spinal Cord Injury Quality of Life (SCI-QOL) Resilience-Short Form | 28 weeks
  10-items assessing state resilience; rated from 1-5 (never-always); score range from 19-50, higher score = more resilient /better outcome
Patient Health Questionnaire-9 | 0 weeks
  9-item depression measure; rated from 0-3 (not at all-nearly every day); score range from 0-27, higher scores = more depressed /worse outcome
Patient Health Questionnaire-9 | 8 weeks
  9-item depression measure; rated from 0-3 (not at all-nearly every day); score range from 0-27, higher scores = more depressed /worse outcome
Patient Health Questionnaire-9 | 16 weeks
  9-item depression measure; rated from 0-3 (not at all-nearly every day); score range from 0-27, higher scores = more depressed /worse outcome
Patient Health Questionnaire-9 | 28 weeks
  9-item depression measure; rated from 0-3 (not at all-nearly every day); score range from 0-27, higher scores = more depressed /worse outcome
Spinal Cord Injury Quality of Life (SCI-QOL) Positive Affect and Wellbeing | 0 weeks
  10-items assessing aspects of well-being; rated from 1-5 (never-always); score range from 10-50, higher score = greater well-being /better outcome
Spinal Cord Injury Quality of Life (SCI-QOL) Positive Affect and Wellbeing | 8 weeks
  10-items assessing aspects of well-being; rated from 1-5 (never-always); score range from 10-50, higher score = greater well-being /better outcome
Spinal Cord Injury Quality of Life (SCI-QOL) Positive Affect and Wellbeing | 16 weeks
  10-items assessing aspects of well-being; rated from 1-5 (never-always); score range from 10-50, higher score = greater well-being /better outcome
Spinal Cord Injury Quality of Life (SCI-QOL) Positive Affect and Wellbeing | 28 weeks
  10-items assessing aspects of well-being; rated from 1-5 (never-always); score range from 10-50, higher score = greater well-being /better outcome
Revised Dyadic Adjustment Scale | 0 weeks
  14-items assessing couple satisfaction and how each partner within the couple perceives their relationship; rated on a scale from 0-5; score range from 0-70, higher scores = better adjustment/greater relationship satisfaction /better outcome
Revised Dyadic Adjustment Scale | 8 weeks
  14-items assessing couple satisfaction and how each partner within the couple perceives their relationship; rated on a scale from 0-5; score range from 0-70, higher scores = better adjustment/greater relationship satisfaction /better outcome
Revised Dyadic Adjustment Scale | 16 weeks
  14-items assessing couple satisfaction and how each partner within the couple perceives their relationship; rated on a scale from 0-5; score range from 0-70, higher scores = better adjustment/greater relationship satisfaction /better outcome
Revised Dyadic Adjustment Scale | 28 weeks
  14-items assessing couple satisfaction and how each partner within the couple perceives their relationship; rated on a scale from 0-5; score range from 0-70, higher scores = better adjustment/greater relationship satisfaction /better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra L Terrill, PhD, Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - University of Utah, Salt Lake City, Utah
  - McGuire Research Institute, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No